CLINICAL TRIAL: NCT06753071
Title: The Efficacy of Pyridostigmine Therapy After Transurethral Resection of Prostate in Cases with Underactive Urinary Bladder: Prospective Randomized Trial
Brief Title: The Efficacy of Pyridostigmine Therapy After Transurethral Resection of Prostate in Cases with Underactive Urinary Bladder.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ammar Fathi Mohamed AlOrabi, Doctor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pyridostigmine therapy
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Underactive Bladder; TURP(transurethral Resection of Prostate); BPH (Benign Prostatic Hyperplasia)
Keywords: BPH; TURP; underactive bladder; pyridostigmine
MeSH Terms: conditions — Urinary Bladder, Underactive; Prostatic Hyperplasia | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pyridostigmine group (Active Comparator): this group will receive pyridostigmine 60 mg twice daily.
  Interventions: Drug: Pyridostigmine oral tablet
- Control group (Placebo Comparator): This will receive placebo postoperatively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridostigmine oral tablet — Pyridostigmine oral tablet, 60 mg, twice daily, for 3 months
  Arms: Pyridostigmine group
Drug: Placebo — Placebo oral tablet, twice daily, for 3 months
  Arms: Control group

SUMMARY:
The efficacy of pyridostigmine therapy after transurethral resection of prostate in cases with underactive urinary bladder

DETAILED DESCRIPTION:
Underactive bladder is a decrease in detrusor contraction and/or shortening of the contraction time, resulting in an incomplete and/or prolongation of the bladder emptying within the normal time frame. Prolonged bladder outlet obstruction due to prostatic enlargment one of the main causes of bladder hypocontractility. To make a diagnosis, it is necessary to perform a pressure-flow study. Decrease in maximum urine flow rate related to bladder outlet obstruction or poor contractility can be distinguished by pressure-flow study.

parasympathomimetics (cholinergic receptor stimulating agents) could be beneficial for patients with underactive bladder. However, no systematic review with meta-analysis addressing potential benefits or adverse effects exists. Pyridostigmine is a medication used to treat myasthenia gravis and underactive bladder as well.

Patients with underactive bladder after transurethral resection of prostate may still complain of recurrent attacks of obstructive lower urinary tract symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are not younger than 45 or older than 75 years.
* Patients with benign prostatic hyperplasia who are eligible for transurethral resection of prostate.
* Patients who has decreased bladder contractility confirmed by urodynamic study (pressure flow study) and plotted on international continence society (ICS) nomogram.

Exclusion Criteria:

* Patients younger than 45 or older than 75 years.
* Patients who have diabetes.
* Patients with a history of neurological diseases.
* patients with a previous history of pelvic surgery.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Severity of lower urinary tract symptoms | 1, 2 , 3 months postoperative
  Severity of lower urinary tract symptoms will be assessed by International Prostate Symptom Score (IPSS) and expressed in number. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Maximum urine flow rate | 1, 2 , 3 months postoperative
  Maximum urine flow rate will be assessed by flowmetry and measured by milliliter per second.
Post-void residual volume | 1, 2 , 3 months postoperative
  Post-void residual volume will be assessed by ultrasound assessment and measured by centimeter cubic.
Bladder contractility evaluation | 1, 2 , 3 months postoperative
  Bladder contractility will be assessed by urodynamic study. Contractility index is expressed in numbers as follows: strong > 150, normal 100-150, and weak < 100.
Bladder detrusor pressure assessment | 1, 2 , 3 months postoperative
  Bladder detrusor pressure will be assessed by urodynamic study and detrusor pressure measured by CmH2O.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shebin El-Kom, Menoufia, Egypt